CLINICAL TRIAL: NCT01962688
Title: A Randomized Study of Pocket Ultrasound Derived IVC Diameter for Guided Management of Heart Failure
Brief Title: Handheld Ultrasound Evaluation of the Inferior Vena Cava to Guide Heart Failure Treatment
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low enrollment
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Jagat Narula, Associate Dean for Global Affairs, Professor Medicine, Cardiology, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GCO 13-0324; IF1486768 (Other: Mount Sinai)
Record Dates: First submitted 2013-10-10; First posted 2013-10-14 (Estimated); Results first posted 2018-06-06 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Heart Failure
Keywords: Heart Failure; Handheld ultrasound; Inferior Vena Cava
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Handheld ultrasound - inpatient (Experimental): Handheld Ultrasound IVC Diameter Guided Diuretic Therapy Handheld ultrasound of the IVC diameter is used to guide diuretic therapy
  Interventions: Device: Handheld ultrasound
- Sham ultrasound - inpatient (Sham Comparator): Conventional Symptom Guided Diuretic Therapy conventional clinical care as would occur outside of the study. These patients receive a sham ultrasound to facilitate blinding
  Interventions: Device: Sham ultrasound
- Handheld ultrasound - ambulatory (Experimental): Handheld Ultrasound IVC Diameter Guided Diuretic Therapy Handheld ultrasound of the IVC diameter is used to guide diuretic therapy in the ambulatory setting during normal clinic visits.
  Interventions: Device: Handheld ultrasound
- Sham ultrasound - ambulatory (Sham Comparator): Conventional Symptom Guided Diuretic Therapy conventional clinical care as would occur outside of the study. These patients receive a sham ultrasound to facilitate blinding in the ambulatory setting during normal clinic visits.
  Interventions: Device: Sham ultrasound

INTERVENTIONS:
Device: Handheld ultrasound — Handheld ultrasound determination of IVC diameter
  Other Names: VSCAN; Handheld Ultrasound IVC Diameter Guided Diuretic Therapy
  Arms: Handheld ultrasound - ambulatory; Handheld ultrasound - inpatient
Device: Sham ultrasound — sham ultrasound to facilitate blinding
  Other Names: Conventional Symptom Guided Diuretic Therapy
  Arms: Sham ultrasound - ambulatory; Sham ultrasound - inpatient

SUMMARY:
The purpose of this study is to see if using a portable handheld ultrasound to guide diuretic therapy for heart failure patients will prevent hospital readmissions. This study will use a handheld ultrasound called a Vscan to look at a large vessel in the body called the Inferior Vena Cava (a vein leading to your heart) . The study aims to see whether changing diuretic therapy based on the size of this vessel will result in the less hospitalizations for heart failure patients as compared to just symptom guided therapy. This study is composed of two independent non-interacting trials-one in the outpatient setting and one in the inpatient setting.

DETAILED DESCRIPTION:
The purpose of this research study is to investigate the use of pocket ultrasound device, called Vscan, in guiding diuretic therapy in ambulatory and inpatient Congestive Heart Failure (CHF) patients. Specifically, Vscan will be used to monitor Inferior Vena Cava (IVC) diameters with the goal of reaching a 50% reduction in IVC when compared to baseline measurements. We hypothesize that compared to the conventional clinical assessment Guided Diuretic Therapy, this new proposed Vscan guided therapy will result in reduction in hospitalization rates. This study is composed of two independent non-interacting randomized single blinded trials-one in the outpatient setting and one in the inpatient setting. 138 total patients and 300 patients will be recruited to the ambulatory trial and inpatient trial respectively.

1. Objectives The objective of the study is to determine whether a simple one step protocol of increasing diuretics to guide a 50% reduction of IVC diameter from baseline measurements results in reduction in hospitalization rates as compared to those seen in therapy determined on the basis of conventional clinical evaluation by a CHF specialist.
2. Background Congestive heart failure (CHF) remains a leading cause of death in industrialized countries. Despite advances in medical treatment, an estimated 250,000-300,000 CHF patients are hospitalized in the United States each year for symptoms caused by low cardiac output (CO). Although the events that cause acute decompensation are multifactorial, the common pathway associated with decreased ventricular function are autonomic dysfunction and fluid retention. It has been previously suggested that an estimated 50%-66% of CHF hospitalizations may be preventable with improved monitoring of fluid volume status. The size and shape of the inferior vena cava (IVC) is correlated to the central venous pressure and circulating blood volume. Therefore evaluation of the IVC provides an instantaneous non-invasive measure of volume status.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of congestive heart failure
* NYHA class II-IV (ambulatory only)
* left ventricular systolic dysfunction with ejection fraction (EF) < 50%
* history of hospitalization for heart failure within the last year (ambulatory only)
* age >18 years old
* admission to heart failure service (inpatient arm only)

Exclusion Criteria:

* Patients with dyspnea not mainly due to heart failure
* valvular disease requiring surgery
* acute coronary syndromes within the previous 10 days
* revascularization within the previous month
* body mass index higher than 35
* serum creatinine level higher than 2.49 mg/dL
* a life expectancy of less than 3 years from noncardiovascular diseases (ambulatory arm only)
* a life expectancy of less than 1 year from noncardiovascular disease (inpatient arm only)
* non-cardiovascular causes of acute renal failure present on admission that preclude the use of diuretics (inpatient arm only)
* unable to give informed consent
* no follow-up possible
* participating in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2013-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jagat Narula, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lloyd-Jones D, Adams RJ, Brown TM, Carnethon M, Dai S, De Simone G, Ferguson TB, Ford E, Furie K, Gillespie C, Go A, Greenlund K, Haase N, Hailpern S, Ho PM, Howard V, Kissela B, Kittner S, Lackland D, Lisabeth L, Marelli A, McDermott MM, Meigs J, Mozaffarian D, Mussolino M, Nichol G, Roger VL, Rosamond W, Sacco R, Sorlie P, Stafford R, Thom T, Wasserthiel-Smoller S, Wong ND, Wylie-Rosett J; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Executive summary: heart disease and stroke statistics--2010 update: a report from the American Heart Association. Circulation. 2010 Feb 23;121(7):948-54. doi: 10.1161/CIRCULATIONAHA.109.192666. No abstract available. PMID 20177011
- [Background] Solomon SD, Dobson J, Pocock S, Skali H, McMurray JJ, Granger CB, Yusuf S, Swedberg K, Young JB, Michelson EL, Pfeffer MA; Candesartan in Heart failure: Assessment of Reduction in Mortality and morbidity (CHARM) Investigators. Influence of nonfatal hospitalization for heart failure on subsequent mortality in patients with chronic heart failure. Circulation. 2007 Sep 25;116(13):1482-7. doi: 10.1161/CIRCULATIONAHA.107.696906. Epub 2007 Aug 27. PMID 17724259
- [Background] O'Connor CM, Abraham WT, Albert NM, Clare R, Gattis Stough W, Gheorghiade M, Greenberg BH, Yancy CW, Young JB, Fonarow GC. Predictors of mortality after discharge in patients hospitalized with heart failure: an analysis from the Organized Program to Initiate Lifesaving Treatment in Hospitalized Patients with Heart Failure (OPTIMIZE-HF). Am Heart J. 2008 Oct;156(4):662-73. doi: 10.1016/j.ahj.2008.04.030. PMID 18926148
- [Background] Gheorghiade M, Filippatos G, De Luca L, Burnett J. Congestion in acute heart failure syndromes: an essential target of evaluation and treatment. Am J Med. 2006 Dec;119(12 Suppl 1):S3-S10. doi: 10.1016/j.amjmed.2006.09.011. PMID 17113398
- [Background] Drazner MH, Hellkamp AS, Leier CV, Shah MR, Miller LW, Russell SD, Young JB, Califf RM, Nohria A. Value of clinician assessment of hemodynamics in advanced heart failure: the ESCAPE trial. Circ Heart Fail. 2008 Sep;1(3):170-7. doi: 10.1161/CIRCHEARTFAILURE.108.769778. PMID 19675681
- [Background] Januzzi JL Jr, Camargo CA, Anwaruddin S, Baggish AL, Chen AA, Krauser DG, Tung R, Cameron R, Nagurney JT, Chae CU, Lloyd-Jones DM, Brown DF, Foran-Melanson S, Sluss PM, Lee-Lewandrowski E, Lewandrowski KB. The N-terminal Pro-BNP investigation of dyspnea in the emergency department (PRIDE) study. Am J Cardiol. 2005 Apr 15;95(8):948-54. doi: 10.1016/j.amjcard.2004.12.032. PMID 15820160
- [Background] Ommen SR, Nishimura RA, Appleton CP, Miller FA, Oh JK, Redfield MM, Tajik AJ. Clinical utility of Doppler echocardiography and tissue Doppler imaging in the estimation of left ventricular filling pressures: A comparative simultaneous Doppler-catheterization study. Circulation. 2000 Oct 10;102(15):1788-94. doi: 10.1161/01.cir.102.15.1788. PMID 11023933
- [Background] Kircher BJ, Himelman RB, Schiller NB. Noninvasive estimation of right atrial pressure from the inspiratory collapse of the inferior vena cava. Am J Cardiol. 1990 Aug 15;66(4):493-6. doi: 10.1016/0002-9149(90)90711-9. PMID 2386120
- [Background] Blair JE, Brennan JM, Goonewardena SN, Shah D, Vasaiwala S, Spencer KT. Usefulness of hand-carried ultrasound to predict elevated left ventricular filling pressure. Am J Cardiol. 2009 Jan 15;103(2):246-7. doi: 10.1016/j.amjcard.2008.08.061. Epub 2008 Oct 30. PMID 19121445
- [Background] Lucas C, Johnson W, Hamilton MA, Fonarow GC, Woo MA, Flavell CM, Creaser JA, Stevenson LW. Freedom from congestion predicts good survival despite previous class IV symptoms of heart failure. Am Heart J. 2000 Dec;140(6):840-7. doi: 10.1067/mhj.2000.110933. PMID 11099986
- [Background] Gheorghiade M, Follath F, Ponikowski P, Barsuk JH, Blair JE, Cleland JG, Dickstein K, Drazner MH, Fonarow GC, Jaarsma T, Jondeau G, Sendon JL, Mebazaa A, Metra M, Nieminen M, Pang PS, Seferovic P, Stevenson LW, van Veldhuisen DJ, Zannad F, Anker SD, Rhodes A, McMurray JJ, Filippatos G; European Society of Cardiology; European Society of Intensive Care Medicine. Assessing and grading congestion in acute heart failure: a scientific statement from the acute heart failure committee of the heart failure association of the European Society of Cardiology and endorsed by the European Society of Intensive Care Medicine. Eur J Heart Fail. 2010 May;12(5):423-33. doi: 10.1093/eurjhf/hfq045. Epub 2010 Mar 30. PMID 20354029
- [Background] Goonewardena SN, Blair JE, Manuchehry A, Brennan JM, Keller M, Reeves R, Price A, Spencer KT, Puthumana J, Gheorghiade M. Use of hand carried ultrasound, B-type natriuretic peptide, and clinical assessment in identifying abnormal left ventricular filling pressures in patients referred for right heart catheterization. J Card Fail. 2010 Jan;16(1):69-75. doi: 10.1016/j.cardfail.2009.08.004. Epub 2009 Sep 26. PMID 20123321
- [Background] Patel AR, Alsheikh-Ali AA, Mukherjee J, Evangelista A, Quraini D, Ordway LJ, Kuvin JT, Denofrio D, Pandian NG. 3D echocardiography to evaluate right atrial pressure in acutely decompensated heart failure correlation with invasive hemodynamics. JACC Cardiovasc Imaging. 2011 Sep;4(9):938-45. doi: 10.1016/j.jcmg.2011.05.006. PMID 21920330
- [Background] Blehar DJ, Dickman E, Gaspari R. Identification of congestive heart failure via respiratory variation of inferior vena cava diameter. Am J Emerg Med. 2009 Jan;27(1):71-75. doi: 10.1016/j.ajem.2008.01.002. PMID 19041537
- [Background] Hollerbach S, Schultze K, Muscholl M, Scholmerich J. [Ultrasonography of the inferior vena cava (IVC) in the diagnosis and monitoring of therapy in patients with chronic congestive heart failure]. Dtsch Med Wochenschr. 2001 Feb 9;126(6):129-33. doi: 10.1055/s-2001-11047. German. PMID 11233879
- [Background] Guiotto G, Masarone M, Paladino F, Ruggiero E, Scott S, Verde S, Schiraldi F. Inferior vena cava collapsibility to guide fluid removal in slow continuous ultrafiltration: a pilot study. Intensive Care Med. 2010 Apr;36(4):692-6. doi: 10.1007/s00134-009-1745-4. Epub 2010 Jan 22. PMID 20094880
- [Background] Goonewardena SN, Gemignani A, Ronan A, Vasaiwala S, Blair J, Brennan JM, Shah DP, Spencer KT. Comparison of hand-carried ultrasound assessment of the inferior vena cava and N-terminal pro-brain natriuretic peptide for predicting readmission after hospitalization for acute decompensated heart failure. JACC Cardiovasc Imaging. 2008 Sep;1(5):595-601. doi: 10.1016/j.jcmg.2008.06.005. PMID 19356487
- [Background] Gackowski A, Isnard R, Golmard JL, Pousset F, Carayon A, Montalescot G, Hulot JS, Thomas D, Piwowarska W, Komajda M. Comparison of echocardiography and plasma B-type natriuretic peptide for monitoring the response to treatment in acute heart failure. Eur Heart J. 2004 Oct;25(20):1788-96. doi: 10.1016/j.ehj.2004.07.038. PMID 15474693
- [Background] Moreno FL, Hagan AD, Holmen JR, Pryor TA, Strickland RD, Castle CH. Evaluation of size and dynamics of the inferior vena cava as an index of right-sided cardiac function. Am J Cardiol. 1984 Feb 1;53(4):579-85. doi: 10.1016/0002-9149(84)90034-1. PMID 6695787
- [Background] McCullough PA, Nowak RM, McCord J, Hollander JE, Herrmann HC, Steg PG, Duc P, Westheim A, Omland T, Knudsen CW, Storrow AB, Abraham WT, Lamba S, Wu AH, Perez A, Clopton P, Krishnaswamy P, Kazanegra R, Maisel AS. B-type natriuretic peptide and clinical judgment in emergency diagnosis of heart failure: analysis from Breathing Not Properly (BNP) Multinational Study. Circulation. 2002 Jul 23;106(4):416-22. doi: 10.1161/01.cir.0000025242.79963.4c. PMID 12135939
- [Background] Miller JB, Sen A, Strote SR, Hegg AJ, Farris S, Brackney A, Amponsah D, Mossallam U. Inferior vena cava assessment in the bedside diagnosis of acute heart failure. Am J Emerg Med. 2012 Jun;30(5):778-83. doi: 10.1016/j.ajem.2011.04.008. Epub 2011 Jun 12. PMID 21665408
- [Background] Brennan JM, Blair JE, Goonewardena S, Ronan A, Shah D, Vasaiwala S, Kirkpatrick JN, Spencer KT. Reappraisal of the use of inferior vena cava for estimating right atrial pressure. J Am Soc Echocardiogr. 2007 Jul;20(7):857-61. doi: 10.1016/j.echo.2007.01.005. PMID 17617312
- [Background] Wang CS, FitzGerald JM, Schulzer M, Mak E, Ayas NT. Does this dyspneic patient in the emergency department have congestive heart failure? JAMA. 2005 Oct 19;294(15):1944-56. doi: 10.1001/jama.294.15.1944. PMID 16234501
- [Background] Jardin F, Vieillard-Baron A. Ultrasonographic examination of the venae cavae. Intensive Care Med. 2006 Feb;32(2):203-206. doi: 10.1007/s00134-005-0013-5. Epub 2006 Feb 1. No abstract available. PMID 16450103
- [Background] Nagueh SF, Kopelen HA, Zoghbi WA. Relation of mean right atrial pressure to echocardiographic and Doppler parameters of right atrial and right ventricular function. Circulation. 1996 Mar 15;93(6):1160-9. doi: 10.1161/01.cir.93.6.1160. PMID 8653837

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Heart Failure patients presented at outpatient clinics were prospectively recruited.
Groups:
- Handheld Ultrasound: Patients underwent clinical assessment with additional pocket ultrasound (VScan, GE Healthcare) guided assessment of inferior-vena cava for assessing volume status.
- Clinical Assessment Only: Patients underwent clinical assessment without additional pocket ultrasound guided assessment of inferior-vena cava for assessing volume status.
Period: Overall Study
Arm/Group | Handheld Ultrasound | Clinical Assessment Only
Started | 19 | 18
Completed | 19 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Handheld Ultrasound | Clinical Assessment Only | Total
Number analyzed (Participants) | 19 | 18 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.9 (16.7) | 61.5 (11.7) | 61.2 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 13 | 13 | 26
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.3 (4.7) | 26.4 (5.5) | 26.4 (4.9)
Ischemic Cardiomyopathy [Number; unit: participants]
  yes | 8 | 11 | 19
  no | 11 | 7 | 18
Ejection Fraction [Mean (Standard Deviation); unit: percent] | 24.8 (8.4) | 24.2 (9.5) | 24.5 (8.8)
Diuretic use [Number; unit: participants]
  yes | 18 | 15 | 33
  no | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Hospitalized for Cardiovascular Reasons
Description: hospitalization information will be recorded throughout the length of the study for the outpatient arms
Time Frame: up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Handheld Ultrasound | Clinical Assessment Only
Number analyzed (Participants) | 19 | 18
Participants | 4 | 5

2. Primary Outcome: Number of Participants Hospitalized for Non-cardiac Reasons
Description: hospitalization information will be recorded throughout the length of the study for the inpatient arms
Time Frame: up to 6 months
Population: All patients in clinical assessment only group were hospitalized for non-cardiac reasons
Measure: Count of Participants; unit: Participants
Arm/Group | Handheld Ultrasound | Clinical Assessment Only
Number analyzed (Participants) | 19 | 18
Participants | 6 | 18

3. Primary Outcome: Diuretic Change Post-visit
Description: Differences in Changes made in Diuretic doses after Heart failure related visit
Time Frame: 6 months followup
Measure: Count of Units; unit: Number of visits
Units Other Than Participants: Number of visits
Arm/Group | Handheld Ultrasound | Clinical Assessment Only
Number analyzed (Participants) | 19 | 18
Number analyzed (Number of visits) | 31 | 65
Number of visits
  Increase | 10 | 7
  Decrease | 6 | 4
  Stay the same | 15 | 54
Statistical Analysis 1: Comparison: Handheld Ultrasound; Test type: Other; p = 0.002, Chi-squared

4. Secondary Outcome: Number of Participants in Each New York Heart Association Class
Description: New York Heart Association (NYHA) Classification Class I - No symptoms and no limitation in ordinary physical activity, e.g. shortness of breath when walking, climbing stairs etc.
  Class II - Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity.
  Class III - Marked limitation in activity due to symptoms, even during less-than-ordinary activity, e.g. walking short distances (20-100m). Comfortable only at rest.
  Class IV - Severe limitations. Experiences symptoms even while at rest. Mostly bedbound patients.
Time Frame: 6 months
Population: Analyzed total 96 visits
Measure: Number; unit: visits
Units Other Than Participants: Number of Visits
Arm/Group | Handheld Ultrasound | Clinical Assessment Only
Number analyzed (Participants) | 19 | 18
Number analyzed (Number of Visits) | 31 | 65
visits
  NYHA Class I | 0 | 1
  NYHA Class II | 9 | 18
  NYHA Class III | 22 | 39
  NYHA Class IV | 0 | 2

5. Secondary Outcome: Change in Health Related Quality of Life
Description: Change in Health related quality of life at 6 months as compared to at 1 month
Time Frame: 1 month and 6 months
Population: Data not collected
Arm/Group | Handheld Ultrasound | Clinical Assessment Only
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Length of Stay
Description: length of stay in the hospital for inpatient arms only
Time Frame: up to 6 months
Population: Data not collected
Arm/Group | Handheld Ultrasound | Clinical Assessment Only
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 6 months
Description: All Cause Mortality All Cause Hospitalization Cardiac Related Hospitalizations Non-Cardiac Related Hospitalization
Arm/Group | Handheld Ultrasound | Clinical Assessment Only
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/18
Serious Adverse Events (participants affected / at risk) | 7/19 | 10/18
Other Adverse Events (participants affected / at risk) | 0/19 | 0/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Handheld Ultrasound (N=19) | Clinical Assessment Only (N=18)
All cause Hospitalization (Cardiac disorders) | 7 (10) | 9 (23)
Cardiac Related Hospitalization (Cardiac disorders) | 4 (4) | 5 (5)
Non Cardiac Hospitalization (Cardiac disorders) | 3 (6) | 4 (18)

LIMITATIONS AND CAVEATS:
This is a pilot study that involved a small sample size. Because of small sample size, randomization was per visit rather than per patient.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes